CLINICAL TRIAL: NCT02984696
Title: Effects of 6 Months of HRT on Total Antioxidant Capacity in Patients Affected by Hypotalamic Amenorrhea
Brief Title: Total Antioxidant Capacity Before and After HRT in Hypotalamic Amenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypotalamic Amenorrhea-01
Record Dates: First submitted 2016-03-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Hypothalamic Amenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hormonal Replace Therapy (Experimental): 1 mg of transdermal estradiol daily and 10mg of oral Medroxyprogesterone acetate from 16th to 24th day of therapy for six months
  Interventions: Drug: 1 mg of transdermal estradiol daily and 10mg of oral MPA

INTERVENTIONS:
Drug: 1 mg of transdermal estradiol daily and 10mg of oral MPA

SUMMARY:
The aim of our study is to investigate the effects of 6 months oh HRT on total anti-oxidant capacity, clinical, endocrine and metabolic features in women affected by hypotalamic amenorrhea. The study group included 20 patients treated with 1 mg of transdermal estradiol daily and 10mg of oral Medroxyprogesterone acetate from 16th to 24th day of therapy for six months. Menstrual pattern, anthropometric parameters, hormonal assays, DXA and bone metabolism parameters are evaluated before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hypotalamic Amenorrhea

Exclusion Criteria:

* diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 gr oral glucose tolerance test)
* hypertension
* significant liver or renal impairment
* other hormonal dysfunction (hypothalamic, pituitary, PCOS, thiroidal or adrenal)
* neoplasms

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Total Anti-oxidant Capacity | 6 Month

SECONDARY OUTCOMES:
Bone Mineral Density | 6 Months
Osteocalcin | 6 Months
Estrogen levels | 6 Months
number of Cycles in 6 months | 6 Months
  n° of menstrual cycle
beta crosslaps | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of Sacred Heart, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided